CLINICAL TRIAL: NCT02558673
Title: Impact of Diet and Gut Microbiota on Trimethylamine-N-oxide Production and Fate in Humans
Brief Title: Trimethylamine-N-oxide Production and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: American Egg Board (Other); National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: OSP 72118
Record Dates: First submitted 2015-09-08; First posted 2015-09-24 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Trimethylamine-N-oxide; Biomarkers; Production; Metabolism; Gut microbiome; Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Egg (Experimental): Study meals were administered in commonly consumed serving sizes (3 hard-boiled eggs) and provided comparable amounts of TMAO dietary precursors. Each meal was served with one cup of water, administered in a single day and separated by a 1-week washout period.
  Interventions: Other: TMAO dietary precursors
- Beef (Experimental): Study meals were administered in commonly consumed serving sizes (6 oz beef [Philly-Gourmet Beef Patties]) and provided comparable amounts of TMAO dietary precursors. Each meal was served with one cup of water, administered in a single day and separated by a 1-week washout period.
  Interventions: Other: TMAO dietary precursors
- Fish (Experimental): Study meals were administered in commonly consumed serving sizes (6 oz fish [cod fillet]) and provided comparable amounts of TMAO dietary precursors. Each meal was served with one cup of water, administered in a single day and separated by a 1-week washout period.
  Interventions: Other: TMAO dietary precursors
- Fruit (Active Comparator): Study meals were administered in commonly consumed serving sizes (2 single-serve packages of Mott's natural applesauce) and provided comparable amounts of control (or active comparator). Each meal was served with one cup of water, administered in a single day and separated by a 1-week washout period. For the fruit control, 50 mg deuterium-labeled methyl-d9-TMAO (d9-TMAO; Cambridge Isotopes) was added to one cup of water for oral consumption to enable the tracing of the metabolic fate of TMAO, and to assess its bioavailability and clearance.
  Interventions: Other: Control (or active comparator)

INTERVENTIONS:
Other: TMAO dietary precursors
  Arms: Beef; Egg; Fish
Other: Control (or active comparator)
  Arms: Fruit

SUMMARY:
The purpose of this study was to understand the production of trimethylamine-N-oxide (TMAO) and its metabolites from dietary precursors found in fish, eggs and beef. In addition, this study traced the fate of supplemental TMAO that has been labeled with deuterium to determine how TMAO is being used in the body.

DETAILED DESCRIPTION:
Trimethylamine-N-oxide (TMAO) is a carbon-containing organic compound formed from dietary precursors including TMAO (high in fish), choline (high in eggs) and carnitine (high in beef). However, TMAO production is highly variable (Zhang AQ et al., 1999), appears to be influenced by genetics (Cashman JR et al., 2001) and gut microbiome (Wang Z et al., 2011; Koeth RA et al., 2013), and is linked to heart disease in cardiac patients (Wang Z et al., 2011) and colorectal cancer among post-menopausal women (Bae S et al., 2015). At present, very little is known about the metabolic fate of TMAO and how it is used within the human body (Bain MA et al., 2005). This study sought to (i) quantify the effects of eggs, beef and fish on TMAO biomarkers in plasma, muscle, urine and stool; (ii) examine the metabolic fate of supplemental TMAO labeled isotopically with deuterium; and (iii) determine whether TMAO production is a function of the gut microbiome.

To accomplish these objectives, a randomized, controlled cross-over study was conducted in healthy male participants (n=40). The study incorporated four arms comprised of study meals representing animal sources of TMAO (egg, beef and fish) along with a fruit control. The study meals were (i) 3 whole hard-boiled eggs; (ii) 6 oz beef (Philly-Gourmet Beef Patties); (iii) 6 oz fish (cod fillet); and (iv) 2 single-serve packages of Mott's natural applesauce. Each meal was served with one cup of water, administered in a single day and separated by a 1-week washout period. For the fruit control, 50 mg deuterium-labeled methyl-d9-TMAO (d9-TMAO; Cambridge Isotopes) was added to one cup of water for oral consumption to enable the tracing of the metabolic fate of TMAO, and to assess its bioavailability and clearance.

Baseline blood sample was obtained by a phlebotomist using a standard venipuncture procedure, and participants collected their baseline urine sample. They also turned in self-collected baseline 24 h urine and stool samples. Following the consumption of the study meal, serial blood samples were collected at 15, 30 min and 1, 2, 4 and 6 h, while urine samples were collected throughout the 6 h study period. At 4.5 h, participants were provided a fixed fruit snack (i.e., applesauce) and water. On the day that participants consumed the d9-TMAO tracer, participants collected their urine throughout the next 24 h and their stool at the next bowel movement. In addition, a subset of this group (n=6) were invited to undergo a muscle biopsy procedure 6 h after the fruit + d9-TMAO tracer consumption.

ELIGIBILITY:
Inclusion Criteria (main study):

* Healthy men of age 21-50 y
* BMI of 20-29.9 kg/m2 who are willing to comply with the study protocol (consumption of study meals and sample collections)

Inclusion Criteria (sub-study involving muscle biopsy):

* Healthy participants who are able to undergo or watch medical procedures

Exclusion Criteria (main study):

* Men over 50 y of age
* BMI ≥ 30 kg/m2
* Women, vegetarians, smokers, individuals with gastrointestinal diseases or complaints, chronic illnesses or other metabolic diseases (including trimethylaminuria), abnormal laboratory values, and those taking nutritional supplements, antibiotics or probiotics within 2 months of recruitment.

Exclusion Criteria (sub-study involving muscle biopsy):

* Men with history of a negative or allergic reaction to local anesthetics
* Tendency toward easy bleeding or bruising, on medications that may increase the chance of bleeding or bruising (e.g., Aspirin, Coumadin, Anti-inflammatories, Plavix)
* Currently on any immunosuppressive medications (e.g., glucocorticoid steroids, chemotherapy), with disease pathologies that would impair the healing process (e.g., diabetes, cancer, keloids, hereditary healing disorders, jaundice, alcoholism, HIV/AIDS)

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
TMAO biomarkers | Assess change from baseline; randomized, controlled, cross-over design with 4 study sessions with 1-week wash-out between visits. Participants were followed for 6 h (egg, beef and fish), and for 6-24 h (fruit + d9-TMAO)
Gut microbiome profile | Baseline

SECONDARY OUTCOMES:
Flavin monooxygenase 3 (FMO3) 472 G>A | Baseline
One-carbon related biomarkers and carnitine | Assess change from baseline; randomized, controlled, cross-over design with 4 study sessions with 1-week wash-out between visits. Participants were followed for 6 h (egg, beef and fish), and for 6-24 h (fruit + d9-TMAO)

CONTACTS AND LOCATIONS:
Overall Officials: Marie A. Caudill, PhD, Principal Investigator — Cornell University
Locations (2):
- United States (2):
  - Gannett Health Services, Cornell University, Ithaca, New York
  - Human Metabolic Research Unit, Cornell University, Ithaca, New York

REFERENCES:
- [Background] Bae S, Ulrich CM, Neuhouser ML, Malysheva O, Bailey LB, Xiao L, Brown EC, Cushing-Haugen KL, Zheng Y, Cheng TY, Miller JW, Green R, Lane DS, Beresford SA, Caudill MA. Plasma choline metabolites and colorectal cancer risk in the Women's Health Initiative Observational Study. Cancer Res. 2014 Dec 15;74(24):7442-52. doi: 10.1158/0008-5472.CAN-14-1835. Epub 2014 Oct 21. PMID 25336191
- [Background] Bain MA, Fornasini G, Evans AM. Trimethylamine: metabolic, pharmacokinetic and safety aspects. Curr Drug Metab. 2005 Jun;6(3):227-40. doi: 10.2174/1389200054021807. PMID 15975041
- [Background] Cashman JR, Zhang J, Leushner J, Braun A. Population distribution of human flavin-containing monooxygenase form 3: gene polymorphisms. Drug Metab Dispos. 2001 Dec;29(12):1629-37. PMID 11717182
- [Background] Koeth RA, Wang Z, Levison BS, Buffa JA, Org E, Sheehy BT, Britt EB, Fu X, Wu Y, Li L, Smith JD, DiDonato JA, Chen J, Li H, Wu GD, Lewis JD, Warrier M, Brown JM, Krauss RM, Tang WH, Bushman FD, Lusis AJ, Hazen SL. Intestinal microbiota metabolism of L-carnitine, a nutrient in red meat, promotes atherosclerosis. Nat Med. 2013 May;19(5):576-85. doi: 10.1038/nm.3145. Epub 2013 Apr 7. PMID 23563705
- [Background] Wang Z, Klipfell E, Bennett BJ, Koeth R, Levison BS, Dugar B, Feldstein AE, Britt EB, Fu X, Chung YM, Wu Y, Schauer P, Smith JD, Allayee H, Tang WH, DiDonato JA, Lusis AJ, Hazen SL. Gut flora metabolism of phosphatidylcholine promotes cardiovascular disease. Nature. 2011 Apr 7;472(7341):57-63. doi: 10.1038/nature09922. PMID 21475195
- [Background] Zhang AQ, Mitchell SC, Smith RL. Dietary precursors of trimethylamine in man: a pilot study. Food Chem Toxicol. 1999 May;37(5):515-20. doi: 10.1016/s0278-6915(99)00028-9. PMID 10456680
- [Derived] Taesuwan S, Cho CE, Malysheva OV, Bender E, King JH, Yan J, Thalacker-Mercer AE, Caudill MA. The metabolic fate of isotopically labeled trimethylamine-N-oxide (TMAO) in humans. J Nutr Biochem. 2017 Jul;45:77-82. doi: 10.1016/j.jnutbio.2017.02.010. Epub 2017 Apr 13. PMID 28433924